CLINICAL TRIAL: NCT02392052
Title: Enhancing Self-Efficacy for Caregivers of Family Members With Spinal Cord Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Craig Hospital (Other)
Responsible Party: Principal Investigator, Cynthia Harrison-Felix, PhD, Director of Research, Craig Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 713234
Record Dates: First submitted 2015-03-12; First posted 2015-03-18 (Estimated); Last update posted 2019-07-23 (Actual); Status verified 2019-07

CONDITIONS: Spinal Cord Injury
Keywords: caregivers
MeSH Terms: conditions — Spinal Cord Injuries | interventions — Waiting Lists

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Reinvention Protocol Participants (Experimental): This group will receive 6 instructor-led 2 hour long didactic presentations regarding 8 key principles of self-efficacy and experiential exercises, including goal setting and problem solving with extensive group discussion. At the end of each session, tasks are assigned to participants to be completed outside the group during the week between sessions. Experiences from these activities and practice implementing the intervention principles will be shared and discussed each week, providing additional opportunities for problem solving and positive feedback.
  Interventions: Behavioral: Reinvention Protocol Participants
- Waitlist Group (Other): This group will include individuals randomized to receive no treatment for the 18 weeks during which the interventional group will receive the active treatment and have their progress tracked.
  Interventions: Behavioral: Wait List

INTERVENTIONS:
Behavioral: Reinvention Protocol Participants — A cognitive behavioral therapy (CBT), to enhance self-efficacy skills for caregivers of family members with SCI, with a focus on changing thinking styles to help people make emotional and behavioral changes.
  Arms: Reinvention Protocol Participants
Behavioral: Wait List — This group will include individuals randomized to receive no treatment for the 18 weeks during which the interventional group will receive the active treatment and have their progress tracked.
  Arms: Waitlist Group

SUMMARY:
Spinal cord injury (SCI) may result in physical deficits that require assistance from others in order to stay healthy and live independently in a community. The assistance provided by caregivers to a family member with SCI often involves a wide range of activities from helping with basic activities, like toileting and bathing, to managing more complex tasks, such as keeping up with household finances, shopping, and transportation. Caregiving puts demands on an individual's ability to cope and deal with day-to-day stresses, and may be influenced by personal beliefs about one's ability to cope with stress. Beliefs about our ability to perform tasks that affect our lives have been termed "self-efficacy". A strong sense of self-efficacy has been shown to positively impact life choices, motivation, quality of functioning, resilience to adversity, and vulnerability to stress and depression. People with low self-efficacy tend to avoid challenges, discontinue tasks that are difficult, and be at risk for more depression and stress, resulting in less satisfaction with life.

This study uses a psychological strategy, called cognitive behavioral therapy (CBT), to enhance self-efficacy skills for caregivers of family members with SCI, with a focus on changing thinking styles to help people make emotional and behavioral changes. The investigators hypothesize that by providing family caregivers with a six week group educational intervention, their self-efficacy skills as well as general life satisfaction can be improved, and minimize depression, stress and anxiety that often accompany the caregiving role. The innovation of the proposed intervention is its integration of positive psychotherapy concepts into structured group CBT to develop optimistic self-efficacy beliefs, strengthen the caregiver's ability to deal with day-to-day stress, and enhance a sense of well-being in the caregiver which, in turn, may benefit the family member with SCI.

DETAILED DESCRIPTION:
Spinal cord injury (SCI) may result in physical limitations such that receiving assistance from others is critical to maintaining health and facilitating full social integration. The assistance ranges from helping with basic daily activities such as bowel and bladder management, hygiene and dressing, to instrumental activities of daily living, including managing household finances, shopping, or transportation. The challenges that accompany a caregiving role may result in a caregiver's inability to balance responsibilities at home and in the workplace. In addition, there is a tendency for caregivers to neglect their own health, which may jeopardize the ability of the person with SCI to obtain the necessary care and support required for optimal independent functioning. Vulnerability and resilience to the ongoing stresses associated with caregiving for a loved one with SCI may be influenced by personal beliefs about the caregiver's capabilities for coping with them. People's belief about their capabilities for successfully performing tasks that affect their lives has been termed "self-efficacy".

For family caregivers of individuals with SCI, self-efficacy beliefs are essential for coping with the stressors that are experienced in the caregiving role. Anxiety, depression, and a sense of "losing" one's own identity are frequently reported by family caregivers. However, there has been relatively little research regarding caregiving in SCI and even fewer treatment options to enhance self-efficacy for these caregivers. The proposed study involves a randomized clinical trial to examine the effect of an intervention specifically designed by and for family caregivers to help improve self-efficacy and reduce emotional distress associated with it. The goal of this project is to test a six-week manualized, cognitive-behaviorally based group educational intervention to improve family caregivers' self-efficacy beliefs and skills, improve their resilience to the ongoing stresses associated with caregiving, and enhance their overall quality of life with the potential added benefit of improving the quality of life for their family members with SCI. Investigators hypothesize that by providing family caregivers with this educational intervention, the intervention can improve their self-efficacy skills as well as general life satisfaction, and minimize depression, stress and anxiety associated with caregiving. The proposed intervention consists of weekly facilitator-led sessions for a total of 6 weeks and includes didactic presentations of 8 key principles, discussion topics and experiential exercises such as goal setting and problem solving with extensive group discussion. At the end of each session, tasks are assigned to participants to be completed outside the group prior to the next meeting. Session content is organized around concepts of identifying and building character strengths, cultivating positive emotion through focusing on gratitude and on the good in one's life, experientially engaging in pleasurable activities, and accomplishing personal goals. The innovation of the proposed intervention lies in its integration of positive psychotherapy concepts into structured group CBT to develop optimistic self-efficacy beliefs, thereby strengthening the caregiver's resilience to emotional distress, enhancing a sense of well-being in the caregiver which, in turn, may benefit the family member with SCI.

ELIGIBILITY:
Inclusion Criteria:

1. Living with a family member with SCI at any level for whom they are the primary caregiver;
2. 18 years of age or older at the time of study enrollment;
3. English speaking in order to complete study measures and participate in group interactions;
4. score of 30 or lower on the GSES; and
5. able to provide informed consent to participate.

Exclusion Criteria:

1. Not providing any amount of assistance to a family member with SCI;
2. not related through marriage or blood to the person with SCI;
3. lives beyond a reasonable commuting distance from Craig Hospital;
4. unable to verbally communicate;
5. unable to attend group sessions;
6. active participation in another formal clinical group or psychological therapy; or
7. have any condition that, in the judgment of the investigators, precludes successful participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2015-11; Primary Completion 2019-04 (Actual); Study Completion 2019-04 (Actual)

PRIMARY OUTCOMES:
Change in General Self-Efficacy Scale scores over an 18week time period | Baseline, 6 weeks, 18 weeks
  The GSES is a questionnaire designed to assess a person's ability to cope with a variety of difficult demands in life.

SECONDARY OUTCOMES:
Change in the Coping Self-Efficacy Scale (CSES) over an 18 week time period | Baseline, 6 weeks, 18 weeks
  The CSES is a questionnaire designed to assess changes in a person's confidence in his/her ability to cope effectively with a variety of challenges or threats.
Change in the Revised Scale for Caregiving Self-Efficacy (RSCSE) over an 18 week time period | Baseline, 6 weeks, 18 weeks
  The RSCSE is a measure of self-efficacy for obtaining respite, responding to disruptive patient behaviors, and controlling upsetting thoughts about caregiving.
The Diener Satisfaction with Life Scale (SWLS) | Baseline, 6 weeks, 18 weeks
  The SWLS will be used to measure global life satisfaction.
Center for Epidemiological Studies Depression Scale (CES-D) | Baseline, 6 weeks, 18 weeks
  The CES-D is a screening instrument used to measure the current level of depressive symptomatology in general or clinical populations.
General Anxiety Disorder 7-item (GAD-7) | Baseline, 6 weeks, 18 weeks
  The GAD-7 is a brief 7 item measure that will be used to assess the severity of general anxiety.

OTHER OUTCOMES:
Exploratory measure - Hair Cortisol | Baseline, 6 weeks, 18 weeks
  Cortisol is a glucocorticoid hormone secreted by the adrenal gland that functions to restore homeostasis following exposure to stress and is commonly used as an objective biomarker of stress. Cortisol has also been explored as a potential biomarker of well-being; lower levels of salivary cortisol have been associated with higher levels of psychological well-being.

CONTACTS AND LOCATIONS:
Locations (1):
- Craig Hospital, Englewood, Colorado, United States